CLINICAL TRIAL: NCT01385553
Title: Randomized Trial of Fathers for Change: An Intervention for Fathers With Co-Occuring Domestic Violence and Substance Abuse
Brief Title: Fathers for Change for Men With Co-occurring Domestic Violence and Substance Abuse
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Carla Stover, Assistant Professor, Yale University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1003006541; 1K23DA023334-01A2 (NIH)
Record Dates: First submitted 2011-06-14; First posted 2011-06-30 (Estimated); Last update posted 2014-02-19 (Estimated); Status verified 2014-02

CONDITIONS: Domestic Violence; Substance Abuse; Parenting
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Individual Drug Counseling (Active Comparator)
  Interventions: Behavioral: Individual Drug Counseling
- Fathers for Change (Experimental)
  Interventions: Behavioral: Fathers for Change

INTERVENTIONS:
Behavioral: Fathers for Change — FATHERS FOR CHANGE comprises 16, 60 minute sessions of treatment utilizing components of three evidence based practices: SADV-Cognitive Behavioral Therapy, Behavioral Couple Therapy and Child-Parent Psychotherapy. The goals of the intervention are: 1) decreased substance abuse and IPV by teaching coping and anger management skills, 2) improved communication and increased problem solving around shared parenting 3) parenting education including child development and the impact of violence on children, 4) discussion of discipline practices and development of behavior modification or positive reinforcement plans, and 5) attachment focused parent-child play sessions to coach fathers in play with their children and process traumatic experiences.
  Other Names: Integrated Father Treatment for Domestic Violence
  Arms: Fathers for Change
Behavioral: Individual Drug Counseling — Individual drug counseling focuses on the symptoms of drug addiction and related areas of impaired functioning and the content and structure of the patient's ongoing recovery program. This model of counseling is time limited and emphasizes behavioral change. It gives the patient coping strategies and tools for recovery and promotes 12-step ideology and participation. The primary goal of addiction counseling is to assist the addict in achieving and maintaining abstinence from addictive chemicals and behaviors. The secondary goal is to help the addict recover from the damage the addiction has caused in his or her life.
  Other Names: IDC
  Arms: Individual Drug Counseling

SUMMARY:
Social service systems rarely acknowledge the status of men as fathers in the conceptualization and delivery of treatment for substance abuse or domestic violence. Although there has been extensive focus on the treatment of mothers who abuse substances, are victims of intimate partner violence (IPV) (defined as physical aggression and/or psychological abuse and control at the hands of an intimate partner), or maltreat their children there has been little consideration of the need for interventions for fathers with histories of co-morbid IPV and substance abuse. It is estimated that between 10 and 17.8 million children are witness to violence in their homes each year. National and regional samples indicate 50-70% of families impacted by IPV and the typically co-occurring substance abuse have children under the age of seven. Large percentages of these men continue to live with or have consistent contact with their young children despite aggression and substance use.

Court mandated treatments for perpetrators of domestic violence have become the norm, however the efficacy of these treatments is questionable and most do not speak to the broader needs of batterers and their families. How batterer's treatments might impact parenting and father-child relationships and the psychosocial functioning of children is vastly understudied and not currently understood. Since batterer treatments are court mandated and require tremendous financial and community resources, the efficacy of these interventions in stopping the cycle of domestic violence and improving the health and well-being of the batterer, his partner and children is crucial. There are currently NO evidence-based treatments that address co-morbid substance abuse and domestic violence perpetration with emphasis on paternal parenting and the father-child relationship. Consequently, the proposed psychotherapy development project will develop and evaluate the potential efficacy of a novel, relational parent intervention for fathers with co-morbid substance abuse and IPV who have young children. The goals of this intervention are to decrease aggression and substance abuse by increasing focus on fathering and an improved father-child relationship.

ELIGIBILITY:
Inclusion Criteria:

1. meet current DSM-IV criteria for substance abuse and who have used a substance within the 60 days prior to screening;
2. have a police reported incident of IPV (pushing, slapping, kicking) within 6 months of referral;
3. have at least one biological child under the age of 7 with whom they reside or have at least weekly visitation.

Exclusion Criteria:

1. Have histories of severe physical violence (e.g. choking, causing hospitalization);
2. Men who have an active NO CONTACT protective order pertaining to their partner or child;
3. Men whose female partners indicate that they do not want the child to participate;
4. If the female partner indicates that she believes her child is afraid of his/her father and will NOT want to participate;
5. Men who are currently in withdrawal from substances and in need of detoxification;
6. Have cognitive impairment or a lifetime history of any psychotic or bipolar disorder; or
7. Are currently suicidal or homicidal.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2011-06; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Decrease in Verbal and Physical Aggression | Baseline (Start of Tx), 4 month follow-up, 7 month follow-up
  Conflict Tactics Scale and the TimeLine Follow-back calendar interview
Decrease in Substance Abuse | weekly for months 1-4, 7 month followup
  urinalysis results and self report
Decrease in Negative Parenting Behavior | baseline, 4 month, 7 month follow-up
  IOWA, Adult child relationship questionnaire, Parental Acceptance Rejection Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Carla S Stover, Ph.D., Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

REFERENCES:
- [Background] Easton CJ, Mandel DL, Hunkele KA, Nich C, Rounsaville BJ, Carroll KM. A cognitive behavioral therapy for alcohol-dependent domestic violence offenders: an integrated substance abuse-domestic violence treatment approach (SADV). Am J Addict. 2007 Jan-Feb;16(1):24-31. doi: 10.1080/10550490601077809. PMID 17364418